CLINICAL TRIAL: NCT00215020
Title: Phase I Evaluation of Urinary Isoprostane Levels in Pediatric Patients With Inflammatory and Non-Inflammatory Gastrointestinal Disease
Brief Title: Evaluation of Urinary Isoprostanes in the Assessment of Children With Inflammatory Bowel Disease
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: Crohn's and Colitis Foundation (Other)
Responsible Party: Principal Investigator, Paul Rufo, Assistant Professor of Pediatrics, Boston Children's Hospital
Other Study IDs: 03-04-060
Record Dates: First submitted 2005-09-15; First posted 2005-09-22 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Inflammatory Bowel Disease; Ulcerative Colitis; Crohn's Disease
Keywords: Isoprostanes
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Specimens stored at -80 in the Center for IBD at Boston Children's Hospital.
Oversight: Data Monitoring Committee: No

SUMMARY:
Isoprostanes are compounds that are produced as a result of oxidative damage to cell membranes. Elevated tissue, serum, and urinary isoprostane levels have been described in a number of inflammatory diseases. The goal of this study is to determine utility of measuring urinary isoprostane levels in pediatric patients with inflammatory and non-inflammatory gastrointestinal disease. Urine samples will be collected from pediatric patients undergoing procedures in the Children's Hospital endoscopy unit. Clinical disease activity will be assessed using a standardized clinical disease activityiIndex. Gross endoscopic and histologic findings will be graded. Previously obtained laboratory studies will also be recorded. Urinary Isoprostane levels will be determined using a commercially available assay. Isoprostane levels will be compared across conditions (IBD vs. non-inflammatory, Crohn's disease vs. ulcerative colitis) and tested for statistical significance. Similarly, disease severity and urinary isoprostane levels will be assessed. The sensitivity, specificity, and positive and negative predictive values of elevated urinary isoprostane levels at discriminating pediatric patients with inflammatory and non-inflammatory gastrointestinal disease will be calculated.

DETAILED DESCRIPTION:
Isoprostanes are compounds produced as a result of oxidative damage to cell membranes. Elevated tissue, serum, and urinary isoprostane levels have been described in a number of inflammatory diseases. The goal of this study is to determine utility of measuring urinary isoprostane levels in pediatric patients with inflammatory and non-inflammatory gastrointestinal disease. Urine samples will be collected from pediatric patients undergoing procedures in the Children's Hospital endoscopy unit. Clinical disease activity will be assessed using a standardized clinical disease activityiIndex. Gross endoscopic and histologic findings will be graded. Previously obtained laboratory studies will also be recorded. Urinary Isoprostane levels will be determined using a commercially available assay. Isoprostane levels will be compared across conditions (IBD vs. non-inflammatory, Crohn's disease vs. ulcerative colitis) and tested for statistical significance. Similarly, disease severity and urinary isoprostane levels will be assessed. The sensitivity, specificity, and positive and negative predictive values of elevated urinary isoprostane levels at discriminating pediatric patients with inflammatory and non-inflammatory gastrointestinal disease will be calculated.

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled for endoscopic evaluation (upper endoscopy, colonoscopy or sigmoidoscopy)
2. Patients currently completing lactose hydrogen breath tests (LHBT)

Exclusion Criteria:

1. Patients with a previous history of HIV and/or chronic Hepatitis (or active acute hepatitis B or C). Patients will be asked about potential blood borne pathogens at the time of enrollment. No additional blood work or serologic testing outside that obtained for routine care will be required for participation in this study.
2. Patients with a documented history of infectious diarrhea (within the past six months): Patients will be asked about previous testing for infectious diarrhea at the time of enrollment. When indicated, subjects will be asked to have primary care providers forward the results of previous testing.
3. Patients with active Reactive Airway Disease (RAD)/Asthma.
4. Patients with heart disease
5. Smokers
6. Patients with Connective tissue diseases (Scleroderma, Lupus, etc)
7. Patients with Renal Disease
8. Subjects must have had recent biochemical studies completed (including CBC, albumin, and ESR) within one month of receipt of sample.

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients with known or suspected IBD.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2003-09; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul A. Rufo, MD, MMSc, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No